CLINICAL TRIAL: NCT03319160
Title: Post-market Clinical Follow-up Study Evaluating the Efficacy and Safety of LifeVest in Real-life Settings in France
Brief Title: LifeVest Safety and Efficacy in Real Life Settings in France
Acronym: WEARIT-FR
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0130
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Sudden Cardiac Death; Left Ventricular Dysfunction; Cardiac Event; Cardiac Arrythmias
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Dysfunction, Left; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- All LifeVest Users: Patients who were prescribed and used a LifeVest in France
  Interventions: Device: Wearable Cardioverter Defibrillator

INTERVENTIONS:
Device: Wearable Cardioverter Defibrillator — A non-invasive wearable cardioverter defibrillator detects and treats VT/VF without the need for bystander intervention
  Other Names: LifeVest

SUMMARY:
This post-market study is a prospective observational study evaluating the efficacy and safety of the LifeVest in real-life settings.

DETAILED DESCRIPTION:
LifeVest has obtained coverage for 4 indications: (i) implantable cardiac defibrillator (ICD) removal due to cardiac device infections, (ii) a bridge to heart transplantation, (iii) in the early post-myocardial infarction period with left ventricular (LV) dysfunction (LVEF <30%), (iv) and a recent coronary revascularization with LV dysfunction (LVEF < 30%). There is no current comparator to LifeVest. In France, patients at high risk for sudden cardiac arrest (SCD) and waiting for heart transplant or ICD are hospitalized or discharged home without any particular ECG monitoring. LifeVest has been demonstrated to automatically detect and terminate rapid ventricular arrhythmias. Introduction of LifeVest into the current patient management would definitely improve the clinical outcomes and benefit the patients with temporary risk of SCD. The use of LifeVest was shown to be effective in protecting patients against SCD in the United States. However, the clinical impact of using LifeVest in France remains unassessed. Therefore we are planning to conduct a post-market study in France to provide efficacy and safety data for the reimbursement dossier renewal before April 2017.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a LifeVest prescription in clinical routine for the following indications:

  1. implantable cardiac defibrillator (ICD) removal due to cardiac device infections,
  2. a bridge to heart transplantation,
  3. in the early post-myocardial infarct (MI) period with left ventricular (LV) dysfunction (LVEF <30%),
  4. a recent coronary revascularization with LV dysfunction (LVEF < 30%).
* Patients who have given their consent to participate.

Exclusion Criteria:

- There are no exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of France All patient who were prescribed a LifeVest were approached for consent. In addition to those prospectively enrolled, patients who had completed LifeVest use prior to the study start were eligible for retrospective enrollment.
Sampling Method: Probability Sample
Enrollment: 1164 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Szymkiewicz, MD, Study Director — Zoll Medical Corporation
Locations (2):
- France (2):
  - Hôpital Européen Georges Pompidou, Paris
  - Clinique PASTEUR, Toulouse

REFERENCES:
- [Derived] Garcia R, Warming PE, Narayanan K, Defaye P, Guedon-Moreau L, Blangy H, Piot O, Leclercq C, Marijon E; WEARIT-France Investigators. Dynamic changes in nocturnal heart rate predict short-term cardiovascular events in patients using the wearable cardioverter-defibrillator: from the WEARIT-France cohort study. Europace. 2023 May 19;25(5):euad062. doi: 10.1093/europace/euad062. PMID 37021342
- [Derived] Garcia R, Combes N, Defaye P, Narayanan K, Guedon-Moreau L, Boveda S, Blangy H, Bouet J, Briand F, Chevalier P, Cottin Y, Da Costa A, Degand B, Deharo JC, Eschalier R, Extramiana F, Goralski M, Guy-Moyat B, Guyomar Y, Hermida JS, Jourda F, Lellouche N, Mahfoud M, Manenti V, Mansourati J, Martin A, Pasquie JL, Ritter P, Rollin A, Tibi T, Yalioua A, Gras D, Sadoul N, Piot O, Leclercq C, Marijon E. Wearable cardioverter-defibrillator in patients with a transient risk of sudden cardiac death: the WEARIT-France cohort study. Europace. 2021 Jan 27;23(1):73-81. doi: 10.1093/europace/euaa268. PMID 33257972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All LifeVest users completing use between May 2014 and December 2016 were approached for retrospective enrollment.
  All patients prescribed a LifeVest January 2017 through March 2018 were approached for prospective enrollment.
  Recruitment took place in France at 88 cardiology centers.
Groups:
- WCD Users: Patients prescribed a wearable cardioverter defibrillator for:
  1. implantable cardiac-defibrillator (ICD) removal due to device infection,
  2. bridge to heart transplantation, or
  3. ischemic cardiomyopathy with left ventricular ejection fraction (LVEF) <30% in the settings of early post-myocardial infarct or after a recent coronary revascularization.
Period: Overall Study
Arm/Group | WCD Users
Started | 1164
Completed | 1157
Not Completed | 7
Not completed — Data not available. | 7

BASELINE CHARACTERISTICS:
Arm/Group | All LifeVest Users
Number analyzed (Participants) | 1157
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183
  Male | 974
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Enrollment type [Count of Participants; unit: Participants]
  Prospective enrollment | 529
  Retrospective enrollment | 628
BMI [Mean (Standard Deviation); unit: kilograms per meter squared] — Body mass index expressed as (weight in kilograms) divided by (height in meters) squared Population: Missing either height or weight information on 21 subjects
  kilograms per meter squared
    number analyzed (Participants) | 1136
    (all) | 26.2 (5.0)
Resting HR [Mean (Standard Deviation); unit: beats per minute] — Resting heart rate as assessed by clinic personnel Population: Missing data on 17 subjects
  beats per minute
    number analyzed (Participants) | 1140
    (all) | 80.0 (17.6)
Indication for use [Count of Participants; unit: Participants] — Indications for use were based on the reimbursement policy of France at the time of the study
  Participants
    ICD extraction due to infection | 119
    Bridge to heart transplant | 88
    Early after myocardial infarction with LVEF 30% or less | 647
    Early after coronary revascularization with LVEF 30% or less | 303
LVEF (4 groups) [Count of Participants; unit: Participants] — Population: Missing data on 8 subjects
  Participants
    >45%: number analyzed (Participants) | 1149
    >45% | 41
    >35% and ≤45%: number analyzed (Participants) | 1149
    >35% and ≤45% | 48
    >25% and ≤35%: number analyzed (Participants) | 1149
    >25% and ≤35% | 483
    ≤25%: number analyzed (Participants) | 1149
    ≤25% | 577
LVEF (3 groups) [Count of Participants; unit: Participants] — Population: Missing data on 8 subjects
  Participants
    ≥35%: number analyzed (Participants) | 1149
    ≥35% | 147
    ≥30% and <35%: number analyzed (Participants) | 1149
    ≥30% and <35% | 251
    <30%: number analyzed (Participants) | 1149
    <30% | 751
NYHA class [Count of Participants; unit: Participants] — Class I: No limitation of physical activity. Class II: Slight limitation of physical activity due to heart failure symptoms. Class III: Marked limitation of physical activity due to heart failure symptoms.
  Class IV: Symptoms of heart failure at rest. Population: Missing information on 360 subjects
  Participants
    Class I: number analyzed (Participants) | 797
    Class I | 140
    Class II: number analyzed (Participants) | 797
    Class II | 320
    Class III: number analyzed (Participants) | 797
    Class III | 238
    Class IV: number analyzed (Participants) | 797
    Class IV | 99

OUTCOME MEASURES:

1. Primary Outcome: Appropriate Shock Events Per Patient
Description: Appropriate shock events were defined as at least one WCD therapy shock delivered during sustained (at least 30 seconds) ventricular tachycardia (VT) or ventricular fibrillation (VF). All shocks delivered within 24 hours of the first shock were considered one event. Adjudication of cardiac rhythms recorded during WCD therapy shocks was performed by 3 cardiologists familiar with device-recorded ECG tracings.
  For assessing incidence per 100 patient years, all appropriate shock events were considered.
Time Frame: start to end of WCD use (3 months typical prescription)
Measure: Count of Participants; unit: Participants
Arm/Group | All LifeVest Users
Number analyzed (Participants) | 1157
Participants
  Patients not shocked for VT or VF | 1139
  Patients with 1 appropriate shock event | 17
  Patients with 2 appropriate shock events | 1
Statistical Analysis 1: Comparison: All LifeVest Users; Test type: Other; Incidence per 100 patient-years = 7.5, 95% CI 2-sided [6.3 to 8.7], Standard Deviation 2.74 — Poisson distribution assumed due to the infrequent nature of the events. Number of appropriate shock events: 19 (17 subjects had one appropriate shock event, one subject had two appropriate shock events). Length of exposure: 253 patient-years

2. Primary Outcome: Risk of Not Receiving Appropriate Shocks When Necessary
Description: While wearing a WCD, how often does a shock not occur when 1) VF or a sustained (> 30 seconds duration) VT occurs and 2) the response buttons are not used. Response button use is a surrogate for either a conscious patient or bystander presence.
Time Frame: from start to end of WCD use (3 months typical prescription)
Population: All recorded occurrences of VF or sustained VT (>30 seconds)
Measure: Count of Units; unit: Recorded instances of VT/VF
Units Other Than Participants: Recorded instances of VT/VF
Groups:
- Subjects With VT/VF: All subjects who had recorded occurrences of VF or sustained VT (>30 seconds)
Arm/Group | Subjects With VT/VF
Number analyzed (Participants) | 36
Number analyzed (Recorded instances of VT/VF) | 42
Recorded instances of VT/VF
  Appropriate shock for VT/VF | 19
  Response buttons used for tolerated VT/VF | 15
  Sustained VT, self-terminated before shock | 8

3. Primary Outcome: Inappropriate Shock Events Per Patient
Description: Inappropriate shock events were defined as having at least one WCD therapy shock delivered when neither sustained (at least 30 seconds in duration) ventricular tachycardia (VT) or ventricular fibrillation (VF) was not present. All shocks delivered within 24 hours of the first shock were considered one event. Adjudication of cardiac rhythms recorded during WCD therapy shocks was performed by 3 cardiologists familiar with device-recorded ECG tracings. For assessing incidence per 100 patient years, all inappropriate shock events were considered.
Time Frame: from start to end of WCD use (3 months typical prescription)
Measure: Count of Participants; unit: Participants
Arm/Group | All LifeVest Users
Number analyzed (Participants) | 1157
Participants
  Patients without inappropriate shock events | 1149
  Patients with 1 inappropriate shock event | 8
Statistical Analysis 1: Comparison: All LifeVest Users; Test type: Other; Incidence per 100 patient-years = 3.2, 95% CI 2-sided [1.9 to 4.4], Standard Deviation 1.78; Poisson distribution assumed due to the infrequent nature of the events. Number of inappropriately shocked events: 8. Length of exposure: 253 patient-years

4. Secondary Outcome: Survival During WCD Use
Description: The number of patients that were alive at the end of the use of the Wearable Cardioverter Defibrillator (WCD) compared to the total population of patients prescribed the LifeVest
Time Frame: from start to end of WCD use (3 months typical prescription)
Measure: Count of Participants; unit: Participants
Arm/Group | All LifeVest Users
Number analyzed (Participants) | 1157
Participants
  Survival to end of prescribed WCD use (WCD wearing period) | 1132
  Death during WCD wearing period | 25
  Death after WCD wearing period | 1

5. Secondary Outcome: Quality of Life Relative to Health State
Description: Measured through the administration of a patient quality of life survey. This survey has been used previously in a published study of patient quality of life.
  Agreement score according to 5-point Likert scale (lower is better):
  1. = Strongly Agree
  2. = Agree
  3. = Neither Agree nor Disagree
  4. = Disagree
  5. = Strongly Disagree
Time Frame: Time of enrollment
Population: Data was collected from prospectively enrolled subjects at selected sites. Not all sites participated in the quality of life surveys.
  Responses were available from 246 of the 529 prospectively enrolled subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prospective Subjects: Data was collected from prospectively enrolled subjects at selected sites.
Arm/Group | Prospective Subjects
Number analyzed (Participants) | 246
units on a scale
  The LifeVest gives me peace of mind: number analyzed (Participants) | 243
  The LifeVest gives me peace of mind | 1.96 (0.9)
  I don't worry as much because I know the LifeVest is protecting me: number analyzed (Participants) | 243
  I don't worry as much because I know the LifeVest is protecting me | 2.17 (1)
  I sleep significantly better knowing I am protected by the LifeVest: number analyzed (Participants) | 242
  I sleep significantly better knowing I am protected by the LifeVest | 2.51 (1.12)
  I feel more confident returning to my normal daily activities when wearing the LifeVest: number analyzed (Participants) | 244
  I feel more confident returning to my normal daily activities when wearing the LifeVest | 2.11 (0.95)
  LifeVest has given me the confidence to perform exercise or cardiac rehabilitation: number analyzed (Participants) | 242
  LifeVest has given me the confidence to perform exercise or cardiac rehabilitation | 2.35 (1.03)
  Wearing the LifeVest makes me take my condition seriously: number analyzed (Participants) | 245
  Wearing the LifeVest makes me take my condition seriously | 1.66 (0.9)
  I take significantly better care of myself since being prescribed the LifeVest: number analyzed (Participants) | 243
  I take significantly better care of myself since being prescribed the LifeVest | 2.14 (1.06)
  I follow lifestyle modification recommendations from my physician | 1.56 (0.68)
  I would recommend LifeVest to family or friends with a similar medical condition | 1.67 (0.9)

6. Other Pre Specified Outcome: Causes of Mortality
Description: Mortality was adjudicated by 3 cardiologists into these categories: Cardiac, Vascular, or Non-cardiovascular.
Time Frame: Duration of prescribed device use, up to 3 months.
Population: Subjects who died during the device prescription period. The prescriptive period ranged from 1 to 3 months.
  One death had no information recorded (retrospective group) and was labeled unknown.
Measure: Count of Participants; unit: Participants
Arm/Group | WCD Users
Number analyzed (Participants) | 25
Participants
  Cardiac cause | 17
  Vascular cause (includes stroke) | 1
  Non-cardiovascular cause | 6
  Unknown (no information available) | 1

7. Other Pre Specified Outcome: Deaths While Wearing the WCD
Description: Deaths during device use (i.e., physically wearing the WCD) were adjudicated by 3 cardiologists as initiated by asystole, initiated by ventricular fibrillation (VF), or having non-arrhythmic causes.
Time Frame: Terminal event may have occurred any time during device use, up to 3 months. All data available up to 24 hours prior to the terminal event was used for adjudication.
Measure: Count of Participants; unit: Participants
Groups:
- Deaths While Wearing the WCD: Any participant who died while wearing the WCD
Arm/Group | Deaths While Wearing the WCD
Number analyzed (Participants) | 9
Participants
  Arrhythmic cause: primary asystole | 0
  Arrhythmic cause: VF (includes electrical storm) | 2
  Non-arrhythmic cause | 7

ADVERSE EVENTS:
Time Frame: Data was collected until the end of the prescribed WCD use time (typically 3 months).
Description: Only serious adverse events considered related to device use were collected. Adverse events were defined as serious if it resulted in life-threatening injury/illness, required medical/surgical intervention to prevent life-threatening injury/illness or permanent impairment, required hospitalization, prolonged a hospital stay, was considered a medically important event, or resulted in death.
Arm/Group | All LifeVest Users
All-Cause Mortality (participants affected / at risk) | 26/1157
Serious Adverse Events (participants affected / at risk) | 6/1157
Other Adverse Events (participants affected / at risk) | 0/1157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All LifeVest Users (N=1157)
Inappropriate shocks (Product Issues) | 4 (4) — Shocked without clinical VT or VF resulting in hospitalization or other medical intervention
Allergy (Skin and subcutaneous tissue disorders) | 1 (1) — An allergy to a constituent of the LifeVest considered as medically important and required hospital stay. This was resolved.
Dyspnea with device alerts (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Paroxysmal dyspnea and LifeVest arrhythmia alerts resulted in hospital admission until resolved.

LIMITATIONS AND CAVEATS:
Observational study. Included retrospective subjects (54%). Multiple criteria for inclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT03319160/Prot_SAP_000.pdf